CLINICAL TRIAL: NCT05341999
Title: Evaluation of the Effect of Cryotherapy Versus Post-operative Ibuprofen Medication on Post-operative Pain in Mandibular Molar Teeth With Symptomatic Irreversible Pulpitis: a Randomized Controlled Trial
Brief Title: Effect of Cryotherapy Versus Post-operative Ibuprofen Medication on Post-operative Pain in Mandibular Molar Teeth With Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yousef Hassan Mohammed Abuhelal, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO3/3/5
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Cryotherapy; Ibuprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Final irrigation with cold saline (cryotherapy). (Experimental): 20ml of 2.5°C cold saline for 5 min
  Interventions: Other: cold saline (cryotherapy)
- Ibuprofen post-operative medication. (Experimental): a single dose of Ibuprofen 400 mg immediately after completion of root canal treatment
  Interventions: Drug: Ibuprofen 400 mg
- Final irrigation with normal saline, and no post-operative medication (Active Comparator): final irrigation will be done using normal saline at room temperature.
  Interventions: Other: Final irrigation with normal saline

INTERVENTIONS:
Other: cold saline (cryotherapy) — using 20ml of 2.5°C cold saline for 5 min
  Arms: Final irrigation with cold saline (cryotherapy).
Drug: Ibuprofen 400 mg — patients will be prescribed ibuprofen medication as a single dose immediately after completion of root canal treatment.
  Arms: Ibuprofen post-operative medication.
Other: Final irrigation with normal saline — final irrigation will be done using normal saline at room temperature.
  Arms: Final irrigation with normal saline, and no post-operative medication

SUMMARY:
Evaluation of the effect of cryotherapy versus post-operative ibuprofen medication on post-operative pain in mandibular molar teeth with symptomatic irreversible pulpitis .

a new technique was proposed to utilize the effect of cold saline on reducing the inflammatory process in the tissue, the so-called cryotherapy.

DETAILED DESCRIPTION:
PICO/

Population: Molar teeth with symptomatic irreversible pulpitis. Intervention I: Final irrigation with cold saline (cryotherapy). Intervention II: Ibuprofen post-operative medication.

Control: Final irrigation with normal saline, and no post-operative medication. Outcome: Post- operative pain.

Sequence of Procedural steps:

1. Full medical and dental history will be obtained from all the patients .
2. Thorough clinical and radiographic examination for the tooth to be treated will be done.
3. The tooth will be anaesthetized and Access cavity will be performed.
4. The canals will be thoroughly irrigated using 3ml syringe of Sodium hypochlorite after every instrument.
5. Canals will be dried using sterile paper points.
6. In the intervention group 1, cryotherapy irrigation will be done using 20ml of 2.5°C cold saline for 5 min, the cold saline will be stored in an icebox with a thermometer calibrated at 2.5°C.
7. In the intervention group 2, the patients will be prescribed ibuprofen medication as a single dose immediately after completion of root canal treatment.
8. In the control group, final irrigation will be done using normal saline at room temperature.
9. Canals will be dried using sterile paper points, and then filled with gutta percha cones corresponding to the same size of the final shaping file and sealed with sealer.
10. The access cavity will then be closed with temporary filling.
11. Post-operative instructions will be given to all patients. • The patient will be asked to rate their pain level according to the given instructions and telecommunication will be scheduled after 3 days to collect the VAS scores and assess the outcome of the treatment. The patients who will be suffered from severe pain, analgesic will be prescribed.

ELIGIBILITY:
Inclusion Criteria: - Patients above 18 years old and to 60.

* Male or female.
* Patients seeking root canal treatment.
* Molar teeth with Symptomatic irreversible pulpitis with preoperative sharp, moderate, or severe pain with normal periapical radiographic appearance or slight widening in lamina dura.
* Systematically healthy patient (ASA I).
* Patient who can understand VAS and sign informed consent.

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders including cardiovascular, respiratory, and gastrointestinal diseases (ASA II, III or IV).
* History of intolerance to NSAIDS.
* Patients with two or more adjacent teeth requiring endodontic treatment.
* External root resorption.
* Internal root resorption.
* Vertical root fracture.
* Periapical lesion.
* Pregnancy.
* Use of ibuprofen in the last 12 hour.
* Bleeding disorder.
* Long term corticosteroid use. 10
* Mobility Grade II or III.
* Pocket depth more than 5mm.
* Previous root canal therapy.
* Non-restorability.
* TMJ problems, bruxism, clenching or traumatic occlusion.
* Inability to perceive the given instructions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 6 hours post-operatively
  The pain will be recorded using the modified visual analogue scale (VAS). • 0, "no pain"
  * 1-3, "mild pain"
  * 4-6, "moderate pain"
  * 7-10, "severe pain" "10" being the most intense pain conceivable.
Post-operative pain | 24 hours post-operatively
  The pain will be recorded using the modified visual analogue scale (VAS). • 0, "no pain"
  * 1-3, "mild pain"
  * 4-6, "moderate pain"
  * 7-10, "severe pain" "10" being the most intense pain conceivable.
Post-operative pain | 48 hours post-operatively
  The pain will be recorded using the modified visual analogue scale (VAS). • 0, "no pain"
  * 1-3, "mild pain"
  * 4-6, "moderate pain"
  * 7-10, "severe pain" "10" being the most intense pain conceivable.